CLINICAL TRIAL: NCT02035072
Title: Phase II Study of Hypofractionated Radio-chemotherapy With Gemcitabine Plus Oxaliplatin for Unresectable Nonmetastatic Locally Advanced Pancreatic Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST157.01; 2010-020379-22 (EudraCT Number)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Unresectable Pancreatic Cancer; Nonmetastatic Pancreatic Cancer; Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypofractionated RT + Gem + Oxali (Experimental): Hypofractionated radiotherapy + Gemcitabine + Oxaliplatin
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Radiation: Hypofractionated RT

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m2
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2
  Other Names: oxalipaltin
Radiation: Hypofractionated RT — Hypofractionated radiotherapy (35 Gy in 7 fractions)

SUMMARY:
Title: Phase II study of hypofractionated radio-chemotherapy with gemcitabine plus oxaliplatin for unresectable nonmetastatic locally advanced pancreatic cancer.

Protocol code: IRST157.01

Phase: II

Study Design: monocentric, prospective, open-label not randomized trial.

Description of Study Treatment: radio-chemotherapy schedule

* GEMOX: Gemcitabine (GEM) 1000 mg/m2, day 1, and Oxaliplatin (OX) 100 mg/m2, day 2, every 2 weeks for 4 cycles.
* Hypofractionated radiotherapy (35 Gy in 7 fractions in 9 consecutive days, one session per day excluding Saturday and Sunday) administered 15 days after the 4th chemotherapy cycle.
* Further 4 cycles of GEMOX, starting 7-15 days after the end of the radiotherapy.

Objectives:

Step A: primary objective = to evaluate the safety of radiotherapy treatment. Secondary objective = the control of IM (internal margin) intra-fraction.

Step B: primary objective = to evaluate the proportion of the resectable patients after radio-chemotherapy. Secondary objectives = overall Response Rate (ORR); safety profile of combinated treatment;overall survival (OS); local progression free survival (LPFS) and progression free survival (PFS).

Statistical Considerations:

Step A:

Assuming that the probability to observe a toxicity involving the radiotherapy treatment discontinuation with the new treatment is less than 20%, 11 patients are to be evaluated for toxicity. If no toxicity involving the radiotherapy treatment discontinuation will be observed in 11 patients, the treatment can be considered safe with a probability > 90%. If 1 toxicity involving the radiotherapy treatment discontinuation will be observed, 7 more patients needs to be recruited. If no further toxicity involving the radiotherapy treatment discontinuation occurs, the treatment could be considered safe with a probability ≥ 90%.

If 2 or more toxicity involving the radiotherapy treatment discontinuation on 11 patients or 2 or more toxicity involving the radiotherapy treatment discontinuation on 18 patients will be observed, the study will be stopped because not safe and another kind of radiotherapy schedule must be designed.

Step B:

If the radiotherapy treatment will be considered no toxic, the study will continue in Step B : the goal of this phase II study is to increase the proportion of resectable patients of at least 15% with the new radio-chemotherapeutic treatment. By using the single-stage design (Gehan EA, J Chron Dis 1961) a total of 40 patients is required to be recruited in 2 years, and a further one-year period of follow-up is requested. If at least 7 patients out of 40 enrolled will be resectable, the hypothesis that the proportion of resectable patients will be less or equal to P1 (P1=the proportion of resectable patients with the new radio-chemotherapeutic treatment) will be refused and the treatment could be considered active.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed diagnosis of pancreatic cancer are candidates for the trial.
2. Stage III disease (AJCC TNM 6th edition, 2002). Inoperable disease, by radiological and surgical evaluation;
3. Age >18 years and ≤75 years.
4. Life expectancy of greater than 12 weeks.
5. ECOG performance status 0-2 (see Appendix A).
6. Presence of at least of one measurable lesion in agreement to RECIST criteria
7. Patients must have normal organ and marrow function as defined below:

   * Leukocytes >3,000/uL
   * Absolute neutrophil count >1,500/uL
   * Platelets >100,000/uL
   * Total bilirubin < 1.5 X ULN
   * AST (SGOT)/ALT (SGPT) <2.5 X ULN
   * Creatinine < 1.5 X ULN
8. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had any chemotherapy or radiotherapy prior to entering the study;
2. Stage IV disease;
3. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
4. Previous malignancy except cervical carcinoma in situ, adequately treated basal cell carcinoma, superficial bladder tumors, or other malignancies curatively treated >5 years before study entry.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine and oxaliplatin or other agents used in the study.
6. Active brain or leptomeningeal disease
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Toxicity | 15 months after the start of recruitment
  If no toxicity in 11 patients, the treatment can be considered safe with a probability > 90%.
  If 1 toxicity will be observed, 7 more patients needs to be recruited. If no further toxicity occurs, the treatment could be considered safe with a probability ≥ 90%.
  If 2 or more toxicity in 11 patients or 2 or more in18 patients will be observed, the study will be stopped because not safe.
Proportion of resectable patients | 3 years after the start of recruitment
  If at least 7 patients out of 40 enrolled will be resectable, the hypothesis that the proportion of resectable patients will be less or equal to P1 (P1=the proportion of resectable patients with the new radio-chemotherapeutic treatment) will be refused and the treatment could be considered active.

SECONDARY OUTCOMES:
Objective tumor response | 3 years after the start of recruitment.
  It is assessed using RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
Objective tumor response rate (ORR) | 3 years after the start of recruitment.
  It is defined as the proportion of the intention-to-treat (ITT) population showing a complete or partial response, if confirmed ≥ 4 weeks later.
Overall survival (OS) | 3 years after the start of recruitment
  It is counted from the date of registration to the date of death due to any cause or last date the patient was known to be alive (censored observation).
Progression free survival (PFS/local PFS) | 3 years after the start of recruitment
  It is counted from the date of registration to the date of the first observation of documentation of objective disease progression/local disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Romeo, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (1):
- Radiotherapy Unit, IRCCS IRST, Meldola, FC, Italy